CLINICAL TRIAL: NCT01492296
Title: Safety, Quality and Comfort of Upper Gastrointestinal Endoscopy With Conscious Sedation After Fasting for Two Hours
Brief Title: Endoscopy With Short Fasting
Acronym: safendoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade de Passo Fundo (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Fernando Fornari, Clinical Professor, Universidade de Passo Fundo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: safendoscopy
Record Dates: First submitted 2011-12-05; First posted 2011-12-14 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Upper Gastrointestinal Symptoms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional fasting (Active Comparator): patients were evaluated after fasting for 8 hours
  Interventions: Procedure: conventional fasting
- Short fasting (Experimental): patients who were evaluated with endoscopy after fasting for two hours
  Interventions: Procedure: endoscopy after short fasting

INTERVENTIONS:
Procedure: endoscopy after short fasting — patients were evaluated with endoscopy after fasting for two hours
  Arms: Short fasting
Procedure: conventional fasting — patients were evaluated after fasting for 8 hours
  Arms: conventional fasting

SUMMARY:
Upper gastrointestinal (GI) endoscopy is widely used in the clinical practice. An empty stomach is required to ensure quality and safety. For this reason, endoscopy is conventionally performed after 8 or more hours of fasting, which is potentially related to discomfort to the patients. In recent studies, surgical cholecystectomy has been described to be safe after two hours of fasting on liquids. The aim of this study is to assess safety, quality and comfort of upper GI endoscopy after two hours of fasting.

ELIGIBILITY:
Inclusion Criteria:

* elective endoscopy

Exclusion Criteria:

* poor clinical condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
safety | 10 min (endoscopy duration)
  safety of endoscopy after fasting for two hours will be assessed by means of a questionnaire replied by the endoscopists, questioning occurrence of aspiration and regurgitation of gastric contents into the esophagus.

SECONDARY OUTCOMES:
quality | 10 min (endoscopy duration)
  Quality of endoscopy will be assessed by means of a questionnaire replied by the endoscopists, including (1) presence of liquid in the gastric lumen (2) quality of mucosa visualization (3)period needed for gastric aspiration
Endoscopy comfort | 8 hours
  Endoscopy comfort will be evaluated by the patients by means of a questionnaire replied after the procedures. It will include questions about thirst, hunger, anxiety, weakness and nausea.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Koeppe AT, Lubini M, Bonadeo NM, Moraes I Jr, Fornari F. Comfort, safety and quality of upper gastrointestinal endoscopy after 2 hours fasting: a randomized controlled trial. BMC Gastroenterol. 2013 Nov 9;13:158. doi: 10.1186/1471-230X-13-158. PMID 24209639